CLINICAL TRIAL: NCT07387289
Title: Eating Fruits and Vegetables With Pleasure! A Pilot Randomized Controlled Feasibility and Acceptability Assessment of a Nutritional Intervention Integrating Eating Pleasure to Promote Healthy Eating in Higher-Weight Adults
Brief Title: Eating Fruits and Vegetables With Pleasure!
Acronym: PLAISIR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Simone Lemieux, Full Professor, Laval University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2025-480; PJT-175185 (Other Grant/Funding Number: Canadian Institutes of Health Research (CIHR))
Record Dates: First submitted 2026-01-19; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Healthy Eating
Keywords: Fruits; Vegetables; Adults; Higher weight; Nutritional intervention; Feasibility study
MeSH Terms: interventions — Vegetables

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Participants receiving a newly developed, 12-week pleasure-oriented intervention that promotes the consumption of fruits and vegetables.
  Interventions: Behavioral: Eating fruits and vegetables with pleasure!
- Control group (No Intervention): Participants receiving no intervention.

INTERVENTIONS:
Behavioral: Eating fruits and vegetables with pleasure! — A newly developed 12-week, pleasure-oriented intervention that promotes the consumption of fruits and vegetables. The program was designed using the Intervention Mapping framework. It includes 10 group sessions along with an individual follow-up throughout the 12-week period.
  Arms: Intervention group

SUMMARY:
The objective of this interventional study is to pilot test a newly evidence-based intervention integrating different dimensions of eating pleasure to promote the consumption of fruits et vegetables. The target population for this study is men and women, aged 18-65 years old, living with a higher weight.The main hypothesis is that this newly pleasure-oriented intervention is feasible and acceptable for the target population. Participants will be randomized in two groups, a first group receiving the newly, 12-week pleasure-oriented intervention (intervention group) and a second group receiving no intervention (control group).

Participants will:

* Complete a battery of online questionnaires at home before and after the 12-week nutritional intervention (both intervention and control groups);
* For participants assigned to the intervention group only: take part in a 12-week nutritional intervention consisting of 10 group sessions held at Laval University (approximately 2 hours each) and an individual follow-up by phone (30 to 45 minutes). After each session, participants will complete a short questionnaire assessing their appreciation of the session (5 to 10 minutes), as well as a comprehensive appreciation questionnaire at the end of the 12-week intervention (25 to 30 minutes).

DETAILED DESCRIPTION:
Research Problem and Hypothesis The health impact of several nutrients, foods, and certain dietary patterns is well documented. Despite this knowledge, food choices within the population remain suboptimal. Furthermore, attempting to promote healthy eating by focusing on the nutritional quality of foods can present certain pitfalls. Indeed, some studies have suggested that there is a persistent perception across different populations-particularly among individuals with higher body weight - that foods considered "healthy" are necessarily less tasty than "unhealthy" foods. This perception may undermine efforts to adhere to healthy eating, given the importance of taste and the pleasure of eating in everyday food choices. In this context, an approach that leverages the pleasure of eating as a driver for healthy eating could be highly relevant. Interestingly, there is growing evidence that eating pleasure can be used to promote healthy eating. Nevertheless, no systematically developed, evidence-based intervention integrating eating pleasure to encourage healthier food choices has yet been described in the literature. To address this gap, the investigators designed an intervention aimed at increasing fruit and vegetable consumption among adults with higher body weight by incorporating eating pleasure into intervention strategies. The research team is now at the stage of assessing its feasibility and acceptability. The choice of this target population (i.e., adults with higher body weight) is based on the fact that these individuals are more likely to seek nutritional advice and benefit from improvements in their dietary intake and behaviors. The main hypothesis is that the proposed intervention will be considered feasible and acceptable by this population.

Objectives and Methodological Approach This intervention was developed using Intervention Mapping, a widely used protocol in behavioral science for designing effective, theory-based, evidence-informed interventions that place the needs and perspectives of the target population at the center of the development process.

In accordance with the Intervention Mapping protocol, four specific objectives were formulated:

1. Assess how the target population adheres to the different dimensions of eating pleasure;
2. Explore dietitians' perspectives on the elements to consider to maximize the relevance, feasibility, and applicability of using eating pleasure to promote healthy eating by conducting in-depth interviews exploring how the different dimensions of eating pleasure are used to encourage healthy eating, the challenges , and the themes and activities that should be integrated into the intervention;
3. Develop the intervention in terms of performance and change objectives, theory-based methods and strategies, and intervention components;
4. Conduct a pilot study of the intervention to assess its feasibility and acceptability. To do so, five indicators of feasibility and acceptability will be evaluated: (1) attrition rate, (2) adherence rate, (3) participation rate, (4) perceived acceptability, and (5) implementation fidelity. Performance and change objectives targeted by the intervention will also be measured to identify effective components and those requiring improvement. Measures related to eating pleasure will also be collected, as eating pleasure is considered a key driver of change in this intervention. Dietary quality will be assessed before and after the intervention, as it is the primary outcome of the planned full-scale randomized controlled trial. Finally, certain eating behaviors will also be measured before and after the intervention to ensure that improvements in dietary intake are accompanied by healthy eating behaviors. Similarly, attitudes and beliefs about weight will be assessed to evaluate the impact of the intervention on these variables.

The present application concerns specific objective 4. The intervention will last 12 weeks and include 10 group sessions as well as an individual follow-up.

Participants and Recruitment A total of 88 participants will be recruited and randomly assigned to one of two study groups: a control group (no intervention, n = 44) and an intervention group (n = 44). Allocation will ensure equitable gender representation, with an equal number of men and women in each group. Participants identifying as "other" gender will also be evenly distributed between the two groups. Half of the participants in each group will be aged 18-42 years, and the other half will be aged 43-65 years (42 years being the median age of the 18-65 population in Quebec).

Inclusion criteria are: (1) aged 18-65 years; (2) presenting with higher body weight, defined in this study as a body mass index (BMI) ≥ 30 kg/m²; (3) able to come to INAF (Laval University) if randomized to the intervention group; and (4) to be fluent in French, as the nutrition intervention will be conducted in this language. Participants without Internet access will be able to come to Laval University to complete their online questionnaires, reducing recruitment bias associated with socioeconomic status. Individuals currently suffering from or with a history of eating disorders (e.g., binge eating disorder, anorexia, or bulimia), as well as pregnant or breastfeeding, will be excluded from this study, as these conditions may significantly influence perceptions related to eating pleasure and healthy eating.

Participants will be recruited through mailing lists of the research institute (INAF) and Laval University (students and staff), as well as via social media (e.g., Facebook, Instagram), the INAF website, and certain community collaborators and affiliated centers of the co-investigators. Interested individuals will be invited to contact the research team and provide their phone number. A team member will then call them to present the study and ask a few questions to assess eligibility. Once eligibility is confirmed, the consent form will be presented via the secure FANI platform. If participants have questions, they will be invited to contact the research team. They will have as much time as needed to consider participation. Those wishing to take part in the study will be asked to indicate their consent in the online consent form.

Randomization Men and women from the two age subgroups described above will be evenly distributed between two groups: one group will receive the intervention, and the other will receive no intervention (control group). It has been suggested that, in pilot studies, a no-treatment control group may be preferable to avoid prematurely discarding a potentially promising intervention. The intervention will be facilitated by one or more dietitians involved in the steering committee responsible for developing the intervention. To minimize bias, the randomization sequence for participants will be generated by a computer algorithm using random numbers, taking into account participants' gender and age.

Steering Committee As recommended in the Intervention Mapping process, a steering committee was established at the beginning of the project to provide support, guidance, and oversight at key stages. This committee includes the researchers and the student involved in the project, three dietitians working with the target population, and two individuals from the target population (one man and one woman).

Statistical Analyses Quantitative data related to feasibility and acceptability measures will be presented as means and percentages. For qualitative data, an inductive thematic content analysis will be conducted independently by two team members using NVivo software. Sociodemographic data (e.g., age, gender, income, education level, ethnicity or cultural background) will be entered as attributes to determine whether they influence expressed feedback.

Changes in dependent variables (HEFI-2019, HEFI-FV, IES-3 and DEBQ scales, performance objectives, eating pleasure scales, FAAT) will be compared between intervention and control groups using the PROC MIXED procedure for repeated measures in SAS software (Cary, NC). Confounding variables (e.g., age, gender, income, education level, ethnicity/cultural background, obesity-related comorbidities) and their interactions with the intervention effect will be tested and included as covariates in the models.

Contribution to Knowledge Advancement This study will make a significant contribution to advancing knowledge in healthy eating promotion by leveraging eating pleasure as an innovative driver. The surveys with individuals with higher body weight and dietitians revealed new ways in which eating pleasure can be used to support healthy eating. This intervention will then systematically determine the best way to integrate these findings and other available evidence into practice by health professionals. This project will also provide a new example of collaboration between researchers, clinicians, and the public in generating knowledge that can be rapidly applied.

Perspectives and Knowledge Mobilization Plan This project will help better understand how to use eating pleasure to promote healthy eating among individuals with higher body weight. It will be followed by a randomized controlled trial to evaluate the intervention's effectiveness. Ultimately, an online training workshop for dietitians could be developed to ensure dissemination and sustainability of the intervention, with complementary research to monitor implementation.

Given the significant intercultural differences in food perceptions, the intervention will need to be adapted if researchers or health professionals wish to use it in populations outside Quebec. To this end, a detailed report on the intervention's development on the Open Science Framework platform will be published, and the intervention manual will be available upon request. Thanks to this methodology used in this study, the intervention can be appropriately adapted using effective strategies.

Finally, new knowledge generated by this project will be disseminated through peer-reviewed scientific publications and conference presentations. As a member of the advisory committee established by Health Canada for developing a tool to measure adherence to Canada's Food Guide recommendations, Dr. Lemieux will use the results of this research to contribute to defining the measurement of the recommendation "Enjoy your food" and, eventually, to developing strategies to promote adherence.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 65 years
* Presenting with higher body weight, defined in this study as a body mass index (BMI) ≥ 30 kg/m²
* Fluent in French, as the nutritional intervention is conducted in this language
* Able to travel to Laval University to take part in the nutritional intervention

Exclusion Criteria:

* Current or past diagnosis of an eating disorder (e.g., binge eating disorder, anorexia nervosa, or bulimia nervosa)
* Pregnant or breastfeeding individuals

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Attrition rate | From enrollment to the end of the 12-week intervention
  The attrition rate, defined as the percentage of participants who do not complete the study, will be calculated in both groups (considered acceptable if below 20%). Reasons for dropout will be documented by the research team to identify potential barriers to participation and the timing of withdrawal.
Adherence rate | At the beginning and at the end of the 12-week intervention
  Adherence rates will be measured by completion of pre- and post-intervention questionnaires in both groups (considered successful if questionnaire completion exceeds 70%). Reasons for non-completion will be documented when applicable.
Participation rate | From enrollment to the end of the 12-week intervention.
  To assess participation rates, attendance at each intervention session will be recorded by the research team in the intervention group (considered successful if attendance exceeds 70%). This rate are calculated at two levels:
  * For each participant (attending at least 70% of sessions on average);
  * For each session (at least 70% of participants present). Attendance trends and reasons for absences will be also documented.
Acceptability | Weekly during the 10 weekly group sessions (Weeks 1-10), and at the individual session conducted at the end of the 12-week intervention (Week 12).
  Regarding acceptability, after each session, participants in the intervention group will complete a questionnaire assessing perceived usefulness and appreciation of the activities (considered acceptable if the average score exceeds 7/10). This questionnaire will also include questions on the understanding of the session content, its credibility, session length, and intention to apply learned concepts. Participants will be invited to indicate what they liked and disliked, suggest improvements, and state whether they would recommend the session to others. At the end of the pilot study, an additional questionnaire will explore overall appreciation of the intervention, including general satisfaction, relevance of the intervention, perceived feasibility of maintaining changes, and willingness to continue or participate in a similar program. Open-ended questions will identify the most liked and disliked aspects, encountered obstacles, and suggested improvements to increase acceptability.
Implementation fidelity | Weekly during the 10 weekly group sessions (Weeks 1-10), and at the individual session conducted at the end of the 12-week intervention (Week 12).
  Implementation fidelity will be assessed by the dietitian facilitating the sessions using a structured observation checklist to document adherence to the protocol, including content delivery, adaptations made and their rationale, and encountered difficulties. Sessions will be recorded so the research team can review them and provide feedback to the dietitian.
Achievement of change objectives targeted by the intervention, assessed using a structured questionnaire | At the end of the 12-week intervention
  The achievement of change objectives identified through the Intervention Mapping process will be assessed using a structured questionnaire developed for this study. The questionnaire includes items reflecting key determinants targeted by the intervention. Participants in both groups will report their level of attainment of each change objective. Each item assesses a specific change objective and will be analyzed individually to inform refinement and optimization of the intervention. In addition, item responses may be aggregated to compute a composite score summarizing overall achievement of the change objectives.
Achievement of intervention performance objectives assessed using a structured questionnaire | At the beginning and at the end of the 12-week intervention
  The achievement of performance objectives identified through the Intervention Mapping process will be assessed using a structured questionnaire developed for this study. The questionnaire includes items reflecting key targeted behavioral objectives addressed by the intervention. Participants in both groups will rate their level of attainment of each performance objective. Each item assesses a specific performance objective and will be analyzed individually to inform refinement and optimization of the intervention. In addition, item responses may be aggregated to compute a composite score summarizing overall achievement of the performance objectives.
Eating pleasure assessed using the Eating Pleasure Questionnaire | At the beginning and at the end of the 12-week intervention
  The Eating Pleasure Questionnaire will be completed to assess whether eating pleasure evolves following participation. This questionnaire will be completed in both groups. Total and subscale scores will be calculated (min:0, max:3), with higher scores indicating greater levels of eating pleasure.
Perceived Impact of Eating Pleasure on Healthy Eating assessed using the Perceived Impact of Eating Pleasure on Healthy Eating questionnaire | At the beginning and at the end of the 12-week intervention
  The Perceived Impact of Eating Pleasure on Healthy Eating questionnaire will be assessed in both groups to assess whether this concept evolves following participation. Total and subscale scores will be calculated (min:1, max:5). A score > 3 indicates that participants perceived eating pleasure as supporting healthy eating, whereas a score < 3 indicated that it is seen as hindering healthy eating.

SECONDARY OUTCOMES:
Diet quality | At the beginning and at the end of the 12-week intervention
  Since this intervention aims to improve participants' dietary quality, the HEFI-2019 score, a global indicator of adherence to the 2019 Canada's Food Guide recommendations, will be measured before and after the intervention in both groups. In addition to the overall score (min:0, max:80), the score for each component will be also calculated to better capture changes in participants' diets. Because the intervention seeks to promote fruit and vegetable consumption, special attention will be given to the fruit and vegetable component (HEFI-FV; min:0, max:20). These scores will be calculated from three validated web-based 24-hour dietary recalls, completed on three unannounced days (two weekdays and one weekend day), randomly selected by a computer algorithm during the week preceding and following the intervention. Higher scores indicate higher diet quality.
Eating behaviors assessed using the Dutch Eating Behavior Questionnaire | At the beginning and at the end of the 12-week intervention
  Participants in both groups will complete the Dutch Eating Behavior Questionnaire (DEBQ), a tool used for measuring restrictive eating, emotional eating, and external eating behaviors. The Dutch Eating Behavior Questionnaire consists of 33 items rated on a 5-point Likert scale (1 = never to 5 = very often). Subscale scores are typically calculated as the mean of their respective items, yielding scores ranging from 1 to 5, with higher scores indicating greater levels of restrained, emotional, or external eating
Attitudes and beliefs about weight | At the beginning and at the end of the 12-week intervention
  Two subscales (" Body acceptance " et " Critical health ") of the Fat Attitudes Assessment Toolkit (FAAT) will be completed by participants in both groups to determine whether attitudes and beliefs about weight influence response to the intervention and whether they change as a result of the intervention. The Body Acceptance and Critical Health subscales of the Fat Attitudes Assessment Toolkit are scored as the mean of their respective items, yielding scores ranging from 1 to 7, with higher scores indicating greater body acceptance and more critical health-related attitudes toward weight.
Intuitive eating behaviors assessed using the Intuitive Eating Scale-3 | At the beginning and at the end of the 12-week intervention
  Participants in both groups will complete the Intuitive Eating Scale-3, a validated questionnaire designed to assess intuitive eating. Items of the Intuitive Eating Scale-3 are rated on a 5-point Likert scale (1 = strongly disagree to 5 = strongly agree). Total and subscale scores (Unconditional Permission to Eat, Eating for Physical Rather than Emotional Reasons, Reliance on Hunger and Satiety Cues, and Body-Food Choice Congruence) are calculated as the mean of their respective items, resulting in scores ranging from 1 to 5, with higher scores indicating greater intuitive eating.

OTHER OUTCOMES:
Sociodemographic Data | At the beginning of the 12-week intervention
  A questionnaire on sociodemographic and medical data-documenting age, gender, income, education level, ethnicity, and obesity-related comorbidities-will be completed by participants prior to the intervention in both groups.

CONTACTS AND LOCATIONS:
Overall Officials: Simone Lemieux, Ph.D., Principal Investigator — Laval University
Locations (1):
- Institut sur la nutrition et les aliments fonctionnels (INAF), Université Laval, Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No
The data underlying the findings are not publicly available because the original approval by the Research Ethics Committee of Laval University and the informed consent from the subjects participating in the studies did not include such a direct, free access. Data can be requested from the principal investigator at simone.lemieux@fsaa.ulaval.ca for researchers who meet the criteria for access to confidential data.

REFERENCES:
- [Background] Cain, P., Donaghue, N., & Ditchburn, G. (2022). Development and validation of the Fat Attitudes Assessment Toolkit (FAAT): A multidimensional nonstigmatizing measure of contemporary attitudes toward fatness and fat people. Journal of Applied Social Psychology, 52, 1121-1145. https://doi.org/10.1111/jasp.12882
- [Background] van Strien, T., Frijters, J. E. R., Bergers, G. P. A., & Defares, P. B. (1986). The Dutch Eating Behavior Questionnaire (DEBQ) for assessment of restrained, emotional, and external eating behavior. International Journal of Eating Disorders, 5(2), 295-315. https://doi.org/10.1002/1098-108X(198602)5:2<295::AID-EAT2260050209>3.0.CO;2-T
- [Background] Tylka TL, Maiano C, Fuller-Tyszkiewicz M, Linardon J, Burnette CB, Todd J, Swami V. The Intuitive Eating Scale-3: Development and psychometric evaluation. Appetite. 2024 Aug 1;199:107407. doi: 10.1016/j.appet.2024.107407. Epub 2024 May 9. PMID 38729580
- [Background] Brassard D, Elvidge Munene LA, St-Pierre S, Gonzalez A, Guenther PM, Jessri M, Vena J, Olstad DL, Vatanparast H, Prowse R, Lemieux S, L'Abbe MR, Garriguet D, Kirkpatrick SI, Lamarche B. Evaluation of the Healthy Eating Food Index (HEFI)-2019 measuring adherence to Canada's Food Guide 2019 recommendations on healthy food choices. Appl Physiol Nutr Metab. 2022 May;47(5):582-594. doi: 10.1139/apnm-2021-0416. Epub 2022 Jan 14. PMID 35030069
- [Background] Brassard D, Elvidge Munene LA, St-Pierre S, Guenther PM, Kirkpatrick SI, Slater J, Lemieux S, Jessri M, Haines J, Prowse R, Olstad DL, Garriguet D, Vena J, Vatanpatast H, L'Abbe MR, Lamarche B. Development of the Healthy Eating Food Index (HEFI)-2019 measuring adherence to Canada's Food Guide 2019 recommendations on healthy food choices. Appl Physiol Nutr Metab. 2022 May;47(5):595-610. doi: 10.1139/apnm-2021-0415. Epub 2022 Jan 14. PMID 35030038
- [Background] Bédard, A., Pitre, C., Grégoire, L.-M., Lévy-Ndejuru, J., Desroches, S., Provencher, V., Bélanger-Gravel, A., Bégin, C., & Lemieux, S. (2025). The Perceived Impact of Eating Pleasure on Healthy Eating: Development and Validation of a Questionnaire for the French-Speaking Québec Adult Population. Dietetics, 4(2), 22. https://doi.org/10.3390/dietetics4020022
- [Background] Gregoire LM, Bedard A, Desroches S, Provencher V, Belanger-Gravel A, Begin C, Lemieux S. Development and validation of a questionnaire assessing eating pleasure dimensions in the adult French-speaking population of the province of Quebec, Canada. Appetite. 2022 May 1;172:105966. doi: 10.1016/j.appet.2022.105966. Epub 2022 Feb 11. PMID 35151684
- [Background] Mohr DC, Spring B, Freedland KE, Beckner V, Arean P, Hollon SD, Ockene J, Kaplan R. The selection and design of control conditions for randomized controlled trials of psychological interventions. Psychother Psychosom. 2009;78(5):275-84. doi: 10.1159/000228248. Epub 2009 Jul 11. PMID 19602916
- [Background] Viechtbauer W, Smits L, Kotz D, Bude L, Spigt M, Serroyen J, Crutzen R. A simple formula for the calculation of sample size in pilot studies. J Clin Epidemiol. 2015 Nov;68(11):1375-9. doi: 10.1016/j.jclinepi.2015.04.014. Epub 2015 Jun 6. PMID 26146089
- [Background] Thabane L, Ma J, Chu R, Cheng J, Ismaila A, Rios LP, Robson R, Thabane M, Giangregorio L, Goldsmith CH. A tutorial on pilot studies: the what, why and how. BMC Med Res Methodol. 2010 Jan 6;10:1. doi: 10.1186/1471-2288-10-1. PMID 20053272
- [Background] Teare MD, Dimairo M, Shephard N, Hayman A, Whitehead A, Walters SJ. Sample size requirements to estimate key design parameters from external pilot randomised controlled trials: a simulation study. Trials. 2014 Jul 3;15:264. doi: 10.1186/1745-6215-15-264. PMID 24993581
- [Background] Statistics Canada (2016). Âge et sexe - Faits saillants en tableaux, Recensement de 2016 [cited October 2 2025]. Available from: https://www12.statcan.gc.ca/census-recensement/2016/dp-pd/hlt-fst/as/index-fra.cfm.
- [Background] Bartholomew Eldredge LK, Markham CM, Ruiter RAC, Fernandez ME, Kok G , Parcel GS. Planning health promotion programs : an intervention mapping approach. San Francisco, CA: Jossey-Bass & Pfeiffer Imprints, Wiley; 2016.
- [Background] Wharton S, Lau DCW, Vallis M, Sharma AM, Biertho L, Campbell-Scherer D, Adamo K, Alberga A, Bell R, Boule N, Boyling E, Brown J, Calam B, Clarke C, Crowshoe L, Divalentino D, Forhan M, Freedhoff Y, Gagner M, Glazer S, Grand C, Green M, Hahn M, Hawa R, Henderson R, Hong D, Hung P, Janssen I, Jacklin K, Johnson-Stoklossa C, Kemp A, Kirk S, Kuk J, Langlois MF, Lear S, McInnes A, Macklin D, Naji L, Manjoo P, Morin MP, Nerenberg K, Patton I, Pedersen S, Pereira L, Piccinini-Vallis H, Poddar M, Poirier P, Prud'homme D, Salas XR, Rueda-Clausen C, Russell-Mayhew S, Shiau J, Sherifali D, Sievenpiper J, Sockalingam S, Taylor V, Toth E, Twells L, Tytus R, Walji S, Walker L, Wicklum S. Obesity in adults: a clinical practice guideline. CMAJ. 2020 Aug 4;192(31):E875-E891. doi: 10.1503/cmaj.191707. No abstract available. PMID 32753461
- [Background] Brown J CC, Johnson Stoklossa C, Sievenpiper J. : Canadian Adult Obesity Clinical Practice Guidelines: Medical Nutrition Therapy in Obesity Management. https://obesitycanada.ca/guidelines/nutrition. Accessed [10/09/2020]. 2020.
- [Background] Jacquier C, Bonthoux F, Baciu M, Ruffieux B. Improving the effectiveness of nutritional information policies: assessment of unconscious pleasure mechanisms involved in food-choice decisions. Nutr Rev. 2012 Feb;70(2):118-31. doi: 10.1111/j.1753-4887.2011.00447.x. PMID 22300598
- [Background] Pettigrew S. Pleasure: An under-utilised 'P' in social marketing for healthy eating. Appetite. 2016 Sep 1;104:60-9. doi: 10.1016/j.appet.2015.10.004. Epub 2015 Oct 9. PMID 26456411
- [Background] Petit O, Merunka D, Anton JL, Nazarian B, Spence C, Cheok AD, Raccah D, Oullier O. Health and Pleasure in Consumers' Dietary Food Choices: Individual Differences in the Brain's Value System. PLoS One. 2016 Jul 18;11(7):e0156333. doi: 10.1371/journal.pone.0156333. eCollection 2016. PMID 27428267
- [Background] Petit, O., Basso, F., Merunka, D., Spence, C., Cheok, A.D. and Oullier, O. (2016), Pleasure and the Control of Food Intake: An Embodied Cognition Approach to Consumer Self-Regulation. Psychol. Mark., 33: 608-619. https://doi.org/10.1002/mar.20903
- [Background] Cornil Y, Chandon P. Pleasure as an ally of healthy eating? Contrasting visceral and Epicurean eating pleasure and their association with portion size preferences and wellbeing. Appetite. 2016 Sep 1;104:52-9. doi: 10.1016/j.appet.2015.08.045. Epub 2015 Sep 10. PMID 26363419
- [Background] Jallinoja P, Pajari P, Absetz P. Negotiated pleasures in health-seeking lifestyles of participants of a health promoting intervention. Health (London). 2010 Mar;14(2):115-30. doi: 10.1177/1363459309353292. PMID 20164161
- [Background] Canadian Foundation for Dietetic Research (2015). Tracking Nutrition Trends 2015 [cited September 1, 2017]. Available from: https://www.cfdr.ca/Sharing/Tracking-Nutrition-Trends.aspx.
- [Background] Raghunathan, R., Naylor, R. W., & Hoyer, W. D. (2006). The Unhealthy = Tasty Intuition and Its Effects on Taste Inferences, Enjoyment, and Choice of Food Products. Journal of Marketing, 70(4), 170-184. https://doi.org/10.1509/jmkg.70.4.170
- [Background] Phan UT, Chambers E 4th. Motivations for choosing various food groups based on individual foods. Appetite. 2016 Oct 1;105:204-11. doi: 10.1016/j.appet.2016.05.031. Epub 2016 May 26. PMID 27235822
- [Background] Dodds A, Chamberlain K. The problematic messages of nutritional discourse: A case-based critical media analysis. Appetite. 2017 Jan 1;108:42-50. doi: 10.1016/j.appet.2016.09.021. Epub 2016 Sep 19. PMID 27659870
- [Background] Demos KE, McCaffery JM, Thomas JG, Mailloux KA, Hare TA, Wing RR. Identifying the mechanisms through which behavioral weight-loss treatment improves food decision-making in obesity. Appetite. 2017 Jul 1;114:93-100. doi: 10.1016/j.appet.2017.03.013. Epub 2017 Mar 15. PMID 28315419
- [Background] Briers B, Huh YE, Chan E, Mukhopadhyay A. The unhealthy = tasty belief is associated with BMI through reduced consumption of vegetables: A cross-national and mediational analysis. Appetite. 2020 Jul 1;150:104639. doi: 10.1016/j.appet.2020.104639. Epub 2020 Feb 22. PMID 32097691
- [Background] Micha R, Penalvo JL, Cudhea F, Imamura F, Rehm CD, Mozaffarian D. Association Between Dietary Factors and Mortality From Heart Disease, Stroke, and Type 2 Diabetes in the United States. JAMA. 2017 Mar 7;317(9):912-924. doi: 10.1001/jama.2017.0947. PMID 28267855
- [Background] Jannasch F, Kroger J, Schulze MB. Dietary Patterns and Type 2 Diabetes: A Systematic Literature Review and Meta-Analysis of Prospective Studies. J Nutr. 2017 Jun;147(6):1174-1182. doi: 10.3945/jn.116.242552. Epub 2017 Apr 19. PMID 28424256
- [Background] Fardet A, Boirie Y. Associations between food and beverage groups and major diet-related chronic diseases: an exhaustive review of pooled/meta-analyses and systematic reviews. Nutr Rev. 2014 Dec;72(12):741-62. doi: 10.1111/nure.12153. Epub 2014 Nov 18. PMID 25406801
- [Background] Sofi F, Macchi C, Abbate R, Gensini GF, Casini A. Mediterranean diet and health status: an updated meta-analysis and a proposal for a literature-based adherence score. Public Health Nutr. 2014 Dec;17(12):2769-82. doi: 10.1017/S1368980013003169. Epub 2013 Nov 29. PMID 24476641
- [Background] Schwingshackl L, Bogensberger B, Hoffmann G. Diet Quality as Assessed by the Healthy Eating Index, Alternate Healthy Eating Index, Dietary Approaches to Stop Hypertension Score, and Health Outcomes: An Updated Systematic Review and Meta-Analysis of Cohort Studies. J Acad Nutr Diet. 2018 Jan;118(1):74-100.e11. doi: 10.1016/j.jand.2017.08.024. Epub 2017 Oct 27. PMID 29111090
- [Background] Mente A, de Koning L, Shannon HS, Anand SS. A systematic review of the evidence supporting a causal link between dietary factors and coronary heart disease. Arch Intern Med. 2009 Apr 13;169(7):659-69. doi: 10.1001/archinternmed.2009.38. PMID 19364995